CLINICAL TRIAL: NCT01151098
Title: An Open-Label, Multi-Center, Titration Study to Establish the Long-term Safety and Tolerability of Buprenorphine Transdermal Delivery System (BTDS) 5 mg, 10 mg, and 20 mg in Patients With Chronic Non-Malignant Pain Syndromes Responsive to Opioid Combination Therapy - a 28-Week Extension Study.
Brief Title: Safety of Buprenorphine Transdermal Systems in Subjects With Chronic Nonmalignant Pain - a 28-week Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUP3201S
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Nonmalignant Pain
Keywords: Chronic nonmalignant pain; Opioid; Transdermal; Butrans (BTDS)
MeSH Terms: interventions — Buprenorphine

ARMS (1):
- BTDS 5, 10 or 20 (Experimental): Buprenorphine transdermal patch
  Interventions: Drug: Buprenorphine transdermal patch

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 5, 10 or 20 mcg/h applied for 7-day wear
  Other Names: Butrans™

SUMMARY:
The objective of this study was to evaluate the long-term safety and tolerability of 7-day BTDS in a 28-week open-label extension phase in subjects with chronic nonmalignant pain syndromes whose pain had been previously controlled by oral opioid combination therapy.

DETAILED DESCRIPTION:
Upon entering the extension phase (BUP3201S), subjects will receive BTDS 5, regardless of their dose level at discontinuation or completion of the BUP3201 core study. Subjects are allowed to titrate after 48 hours to BTDS 10 or 20 that provided stable pain control with minimal tolerability problems. Additional medical therapies are permitted if necessary, and there is no restriction on concomitant analgesic medications. The subjects have weekly visits for 4 consecutive weeks, and every 4 weeks thereafter, until the end of the scheduled extension phase.

ELIGIBILITY:
Inclusion Criteria:

Include:

* Subjects of either sex aged 18 years or older.
* Subjects who have completed or discontinued the double-blind evaluation phase of study BUP3201 are eligible to continue to receive open-label BTDS in the extension.

Exclusion Criteria:

Include:

* Subjects currently receiving daily morphine or oxycodone (mono-therapy).
* Subjects who are discontinued from BUP3201 due to adverse events.
* Subjects who are scheduled for surgery of the disease site (e.g. major joint replacement surgery) or any other major surgery which would fall within the study period.

Refer to core study for additional inclusion/exclusion information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2001-04; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Arizona Research Center Inc., Phoenix, Arizona
  - Clinical Research Consultants Inc, Trumbull, Connecticut
  - Tampa Bay Medical Research Inc, Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - University Clinical Research Deland, DeLand, Florida
  - University Clinical Research Inc,, Pembroke Pines, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - Gold Coast Research LLC, Tamarac, Florida
  - Family Medicine Associates, Evansville, Indiana
  - Pain Management & Rehabilitation, Terre Haute, Indiana
  - Southeastern Center for Headache and Pain, Crestview Heights, Kentucky
  - Westside Family Medical Center PC, Kalamazoo, Michigan
  - The Arthritis Clinic, Charlotte, North Carolina
  - Cornerstone Research Care, High Point, North Carolina
  - ALL-TRIALS Clinical Research LLC, Winston-Salem, North Carolina
  - Summit Research Solutions, Memphis, Tennessee
  - Radiant Research - Austin, Austin, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Clinical Research Management, New Berlin, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16-Apr-2001 (first patient first visit) 27-Feb-2002 (last patient last visit). The extension phase of study was conducted at 20 sites in the US Baseline Period: and 18 sites in the UK.
Pre-assignment Details: Adult subjects aged ≥ 18 years, with chronic nonmalignant pain, controlled on oral opioid therapy. Subjects in the US who participated in the BUP3201 core study and met the criteria per Amendment 2, and subjects in the UK who participated in the BUP3201 core and met the inclusion/ exclusion criteria, were able to participate in the extension.
Groups:
- Total Extension Phase: Buprenorphine transdermal patches (BTDS 5, 10 or 20) applied for 7-day wear.
Period: Overall Study
Arm/Group | Total Extension Phase
Started | 189 (Extension Safety Population)
Completed | 72
Not Completed | 117
Not completed — Adverse Event | 82
Not completed — Lost to Follow-up | 6
Not completed — Lack of Efficacy | 15
Not completed — Protocol Violation | 1
Not completed — Miscellaneous | 13

BASELINE CHARACTERISTICS:
Groups:
- Extension Phase (BTDS 5, 10 or 20): Buprenorphine transdermal patches (BTDS 5, 10 or 20) applied for 7-day wear.
Arm/Group | Extension Phase (BTDS 5, 10 or 20)
Number analyzed (Participants) | 189
Age Continuous [Mean (Standard Deviation); unit: years] | 55.2 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 71
Region of Enrollment [Number; unit: participants]
  United States | 103
  United Kingdom | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) as a Measure of Safety.
Description: Safety was assessed using reports of all new adverse events (AEs) that occurred after the first application of a patch during the extension phase were recorded.
Time Frame: 28 weeks
Population: The Extension Safety population (N = 189) includes all subjects who were exposed to BTDS during the Open-label Extension Phase and provided at least 1 valid safety assessment after exposure to BTDS during the Open-label Extension Phase.
Measure: Number; unit: participants
Groups:
- Total Extension Phase: Buprenorphine transdermal patches (BTDS 5, 10, or 20) applied for 7-day wear.
Arm/Group | Total Extension Phase
Number analyzed (Participants) | 189
participants
  Deaths | 1
  Serious Adverse Events | 16
  All Other Adverse Events in ≥ 4.5% of Subjects | 143

ADVERSE EVENTS:
Time Frame: All adverse events that occurred after administration of the first dose of study drug on or before the final visit were reported and up to 30 days after the end of the trial.
Description: Adverse Events were obtained through spontaneous reports and subject interview.
Arm/Group | Total Extension Phase
Serious Adverse Events (participants affected / at risk) | 16/189
Other Adverse Events (participants affected / at risk) | 143/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Extension Phase (N=189)
Abdominal pain (General disorders) | 1 (1) — Systematic and nonsystematic assessments
Asthenia (General disorders) | 1 (1) — Systematic and nonsystematic assessments
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Systematic and nonsystematic assessments
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Systematic and nonsystematic assessments
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) — Systematic and nonsystematic assessments
Vascular disorder (Vascular disorders) | 2 (2) — Systematic and nonsystematic assessments
Cardiovascular disorder (Cardiac disorders) | 1 (2) — Systematic and nonsystematic assessments
Congestive heart failure (Cardiac disorders) | 1 (1) — Systematic and nonsystematic assessments
Myocardial infarct (Cardiac disorders) | 1 (1) — Systematic and nonsystematic assessments
Peripheral vascular disorder (Vascular disorders) | 1 (1) — Systematic and nonsystematic assessments
Diarrhea (Gastrointestinal disorders) | 1 (1) — Systematic and nonsystematic assessments
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) — Systematic and nonsystematic assessments
Lymphoma-like reaction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Systematic and nonsystematic assessments
Cachexia - Death (Metabolism and nutrition disorders) | 1 (1) — DEATH - Systematic and nonsystematic assessments
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Systematic and nonsystematic assessments
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Systematic and nonsystematic assessments
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (1) — Systematic and nonsystematic assessments
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Systematic and nonsystematic assessments
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Systematic and nonsystematic assessments
Ovarian carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Systematic and nonsystematic assessments
Urinary retention (Renal and urinary disorders) | 1 (1) — Systematic and nonsystematic assessments
Uterine fibroids enlarged (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Systematic and nonsystematic assessments
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Extension Phase (N=189)
Infection (Infections and infestations) | 16 — Systematic and nonsystematic assessments
Pain (General disorders) | 16 — Systematic and nonsystematic assessments
Accidental injury (Injury, poisoning and procedural complications) | 12 — Systematic and nonsystematic assessments
Back pain (General disorders) | 12 — Systematic and nonsystematic assessments
Asthenia (General disorders) | 10 — Systematic and nonsystematic assessments
Constipation (Gastrointestinal disorders) | 13 — Systematic and nonsystematic assessments
Nausea (Gastrointestinal disorders) | 29 — Systematic and nonsystematic assessments
Vomiting (Gastrointestinal disorders) | 13 — Systematic and nonsystematic assessments
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 — Systematic and nonsystematic assessments
Dizziness (Nervous system disorders) | 15 — Systematic and nonsystematic assessments
Somnolence (Nervous system disorders) | 17 — Systematic and nonsystematic assessments
Erythema at site (Skin and subcutaneous tissue disorders) | 61 — Systematic and nonsystematic assessments
Pruritus at site (Skin and subcutaneous tissue disorders) | 42 — Systematic and nonsystematic assessments
Rash at site (Skin and subcutaneous tissue disorders) | 33 — Systematic and nonsystematic assessments
Other site reaction (Skin and subcutaneous tissue disorders) | 17 — Systematic and nonsystematic assessments
Rash (Skin and subcutaneous tissue disorders) | 10 — Systematic and nonsystematic assessments

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days